CLINICAL TRIAL: NCT01564251
Title: An Open-label, Phase I, Dose Escalation Study Evaluating the Safety, Tolerability, and Pharmacokinetics of GDC-0575 Administered Alone and in Combination With Gemcitabine in Patients With Refractory Solid Tumors or Lymphoma
Brief Title: A Study of GDC-0575 Alone and in Combination With Gemcitabine in Participants With Refractory Solid Tumors or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GP28153; 2011-005602-30 (EudraCT Number)
Record Dates: First submitted 2012-03-23; First posted 2012-03-27 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Lymphoma, Solid Tumor
MeSH Terms: conditions — Lymphoma | interventions — GDC-0575; Gemcitabine

ARMS (4):
- Stage 1 Arm 1: GDC-0575 Monotherapy (Experimental): Participants will receive escalating doses of GDC-0575, administered orally, for 3 consecutive days, starting on Days 1, 8, and 15 of each 21-day cycle.
  Interventions: Drug: GDC-0575
- Stage 1 Arm 2a: GDC-0575 + Gemcitabine (750 or 1000 mg/m^2) (Experimental): Participants will receive gemcitabine 750 milligrams per meter square (mg/m^2) or 1000 mg/m^2, intravenously, on Days 1 and 8 followed by escalating doses of GDC-0575 orally, on Days 2 and 9 of each 21-day cycle.
  Interventions: Drug: GDC-0575; Drug: Gemcitabine
- Stage 1 Arm 2b: GDC-0575 plus Gemcitabine (500 mg/m^2) (Experimental): Participants will receive gemcitabine 500 mg/m^2, intravenously, once weekly for approximately 2 consecutive weeks of any 3-week period and escalating doses of GDC-0575 orally approximately 24-hours after each gemcitabine dose.
  Interventions: Drug: GDC-0575; Drug: Gemcitabine
- Stage 2: GDC-0575 plus Gemcitabine (Experimental): Participants will receive GDC-0575 in combination with gemcitabine intravenously (1000 mg/m^2 and/or 500 mg/m^2), at or below the MTDs for the combination treatments that are determined during Stage 1.
  Interventions: Drug: GDC-0575; Drug: Gemcitabine

INTERVENTIONS:
Drug: GDC-0575 — Participants will receive GDC-0575 orally at a starting dose of 15 mg.
  Other Names: RO6845979
Drug: Gemcitabine — Participants will receive gemcitabine intravenously at a dose of 1000 mg/m^2 and/or 500 mg/m^2.
  Other Names: Gemzar
  Arms: Stage 1 Arm 2a: GDC-0575 + Gemcitabine (750 or 1000 mg/m^2); Stage 1 Arm 2b: GDC-0575 plus Gemcitabine (500 mg/m^2); Stage 2: GDC-0575 plus Gemcitabine

SUMMARY:
This open-label, multicenter, Phase I, dose-escalation study will evaluate the safety, tolerability, and pharmacokinetics (PK) of GDC-0575 administered alone or in combination with gemcitabine in participants with refractory solid tumors or lymphoma. In Stage 1, cohorts of participants will receive multiple ascending oral doses of GDC-0575 alone or in combination with intravenous gemcitabine. In Stage 2, participants will receive GDC-0575 orally in combination with intravenous gemcitabine at or below the maximum tolerated dose determined in Stage 1. Anticipated time on study treatment is until disease progression or unacceptable toxicity occurs, up to approximately 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Histologically or cytologically documented, locally advanced or metastatic solid tumors or lymphoma for which standard therapy either does not exist or has proven ineffective or intolerable
* Life expectancy greater than or equal to (>=) 12 weeks, in the opinion of the investigator
* Adequate hematologic, liver, and renal function
* For Stage 2: Participants with human epidermal growth factor receptor 2 (HER2) negative, estrogen-receptor (ER) negative, and progesterone-receptor (PR) negative breast cancer
* For Stage 2: Participants with non-mucinous, platinum-resistant ovarian cancer with documented radiographic progression or relapse according to RECIST within 6 months of receiving platinum-based chemotherapy
* For Stage 2: Participants with histologically or cytologically confirmed diagnosis of squamous non-small cell lung cancer (NSCLC); mixed histology that is predominantly squamous is acceptable

Exclusion Criteria:

* History of prior significant toxicity from a same class of agents as GDC-0575 or gemcitabine requiring discontinuation of treatment
* All acute toxicities related to prior therapy must have resolved prior to study entry, except for alopecia and mild neuropathy
* Current severe, uncontrolled systemic disease (including but not limited to clinically significant cardiovascular, pulmonary, or renal disease or ongoing or active infection) excluding the cancer under study
* History of significant cardiac dysfunction
* History of malabsorption or other condition that would interfere with enteral absorption
* Known human immunodeficiency virus (HIV) infection
* Pregnancy, lactation or breastfeeding
* Known brain metastases that are untreated, symptomatic, or require therapy to control symptoms
* Current use of alpha-adrenergic receptor blockers

For Combination Arm only:

* Any contraindication to gemcitabine therapy
* More than two regimens of cytotoxic chemotherapy for the treatment of locally advanced or metastatic cancer
* History of receiving high-dose chemotherapy requiring bone marrow or stem cell support
* Irradiation to more than 25% of bone marrow-bearing areas

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2012-03-23 (Actual); Primary Completion 2018-01-11 (Actual); Study Completion 2018-01-11 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) | Baseline up to approximately 5 years
Percentage of Participants With Dose-Limiting Toxicities (DLTs) | Stage 1 Arm 1: Day 1 up to Day 21. Stage 1 Arm 2: Day 1 up to Day 22 or 29
Maximum Tolerated Dose (MTD) of GDC-0575 | Stage 1 Arm 1: Day 1 up to Day 21. Stage 1 Arm 2: Day 1 up to Day 22 or 29
Recommended Phase II Dose of GDC-0575 | Stage 1 Arm 1: Day 1 up to Day 21. Stage 1 Arm 2: Day 1 up to Day 22 or 29
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUC0-inf) of GDC-0575 | Stage 1 Arm 1, Cycle 1 of 21 days: predose on Days 1, 2, 3, 8, 15; postdose on Days 1, 2, 3, 4, 5, 8, 15. Stage 1 Arm 2 and Stage 2, Cycle 1 of 21 days: predose and postdose on Days 2, 9 (detailed timeframe is provided in outcome measure description)
  Stage 1 Arm 1, Cycle 1 of 21 days: predose (5 to 30 minutes) on Days 1, 2, 3, 8, 15; 0.5, 1, 1.5, 2, 4, 6, 8 hours (h) postdose on Days 1, 3; 2, 4h postdose on Days 2, 15; 2h postdose on Day 8; on Days 4, 5. Stage 1 Arm 2 and Stage 2, Cycle 1 of 21 days: predose (5 minutes), 0.5, 1, 1.5, 2, 4, 6h postdose on Day 2 (additionally at 8h postdose on Day 2 for Arm 2a only); predose (0.5h), 2h postdose on Day 9
Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) | Stage 1 Arm 1, Cycle 1 of 21 days: predose on Days 1, 2, 3, 8, 15; postdose on Days 1, 2, 3, 4, 5, 8, 15. Stage 1 Arm 2 and Stage 2, Cycle 1 of 21 days: predose and postdose on Days 2, 9 (detailed timeframe is provided in outcome measure description)
  Stage 1 Arm 1, Cycle 1 of 21 days: predose (5 to 30 minutes) on Days 1, 2, 3, 8, 15; 0.5, 1, 1.5, 2, 4, 6, 8 h postdose on Days 1, 3; 2, 4h postdose on Days 2, 15; 2h postdose on Day 8; on Days 4, 5. Stage 1 Arm 2 and Stage 2, Cycle 1 of 21 days: predose (5 minutes), 0.5, 1, 1.5, 2, 4, 6h postdose on Day 2 (additionally at 8h postdose on Day 2 for Arm 2a only) ; predose (0.5h), 2h postdose on Day 9
Maximum Observed Plasma Concentration (Cmax) GDC-0575 | Stage 1 Arm 1, Cycle 1 of 21 days: predose on Days 1, 2, 3, 8, 15; postdose on Days 1, 2, 3, 4, 5, 8, 15. Stage 1 Arm 2 and Stage 2, Cycle 1 of 21 days: predose and postdose on Days 2, 9 (detailed timeframe is provided in outcome measure description)
  Stage 1 Arm 1, Cycle 1 of 21 days: predose (5 to 30 minutes) on Days 1, 2, 3, 8, 15; 0.5, 1, 1.5, 2, 4, 6, 8 h postdose on Days 1, 3; 2, 4h postdose on Days 2, 15; 2h postdose on Day 8; on Days 4, 5. Stage 1 Arm 2 and Stage 2, Cycle 1 of 21 days: predose (5 minutes), 0.5, 1, 1.5, 2, 4, 6h postdose on Day 2 (additionally at 8h postdose on Day 2 for Arm 2a only) ; predose (0.5h), 2h postdose on Day 9
Minimum Observed Plasma Trough Concentration (Cmin) of GDC-0575 | Stage 1 Arm 1, Cycle 1 of 21 days: predose (5 to 30 minutes) on Days 1, 2, 3, 8, 15; Stage 1 Arm 2 and Stage 2, Cycle 1 of 21 days: predose (5 minutes) on Day 2; predose (0.5h) on Day 9
Time to Reach Maximum Observed Plasma Concentration (Tmax) of GDC-0575 | Stage 1 Arm 1, Cycle 1 of 21 days: predose on Days 1, 2, 3, 8, 15; postdose on Days 1, 2, 3, 4, 5, 8, 15. Stage 1 Arm 2 and Stage 2, Cycle 1 of 21 days: predose and postdose on Days 2, 9 (detailed timeframe is provided in outcome measure description)
  Stage 1 Arm 1, Cycle 1 of 21 days: predose (5 to 30 minutes) on Days 1, 2, 3, 8, 15; 0.5, 1, 1.5, 2, 4, 6, 8 h postdose on Days 1, 3; 2, 4h postdose on Days 2, 15; 2h postdose on Day 8; on Days 4, 5. Stage 1 Arm 2 and Stage 2, Cycle 1 of 21 days: predose (5 minutes), 0.5, 1, 1.5, 2, 4, 6h postdose on Day 2 (additionally at 8h postdose on Day 2 for Arm 2a only) ; predose (0.5h), 2h postdose on Day 9
Apparent Terminal Half-Life (t1/2) of GDC-0575 | Stage 1 Arm 1, Cycle 1 of 21 days: predose on Days 1, 2, 3, 8, 15; postdose on Days 1, 2, 3, 4, 5, 8, 15. Stage 1 Arm 2 and Stage 2, Cycle 1 of 21 days: predose and postdose on Days 2, 9 (detailed timeframe is provided in outcome measure description)
  Stage 1 Arm 1, Cycle 1 of 21 days: predose (5 to 30 minutes) on Days 1, 2, 3, 8, 15; 0.5, 1, 1.5, 2, 4, 6, 8 h postdose on Days 1, 3; 2, 4h postdose on Days 2, 15; 2h postdose on Day 8; on Days 4, 5. Stage 1 Arm 2 and Stage 2, Cycle 1 of 21 days: predose (5 minutes), 0.5, 1, 1.5, 2, 4, 6h postdose on Day 2 (additionally at 8h postdose on Day 2 for Arm 2a only) ; predose (0.5h), 2h postdose on Day 9
Apparent Oral Clearance (CL/F) of GDC-0575 | Stage 1 Arm 1, Cycle 1 of 21 days: predose on Days 1, 2, 3, 8, 15; postdose on Days 1, 2, 3, 4, 5, 8, 15. Stage 1 Arm 2 and Stage 2, Cycle 1 of 21 days: predose and postdose on Days 2, 9 (detailed timeframe is provided in outcome measure description)
  Stage 1 Arm 1, Cycle 1 of 21 days: predose (5 to 30 minutes) on Days 1, 2, 3, 8, 15; 0.5, 1, 1.5, 2, 4, 6, 8 h postdose on Days 1, 3; 2, 4h postdose on Days 2, 15; 2h postdose on Day 8; on Days 4, 5. Stage 1 Arm 2 and Stage 2, Cycle 1 of 21 days: predose (5 minutes), 0.5, 1, 1.5, 2, 4, 6h postdose on Day 2 (additionally at 8h postdose on Day 2 for Arm 2a only) ; predose (0.5h), 2h postdose on Day 9
Accumulation Ratio (Rac) of GDC-0575 | Stage 1 Arm 1, Cycle 1 of 21 days: predose on Days 1, 2, 3, 8, 15; postdose on Days 1, 2, 3, 4, 5, 8, 15. Stage 1 Arm 2 and Stage 2, Cycle 1 of 21 days: predose and postdose on Days 2, 9 (detailed timeframe is provided in outcome measure description)
  Stage 1 Arm 1, Cycle 1 of 21 days: predose (5 to 30 minutes) on Days 1, 2, 3, 8, 15; 0.5, 1, 1.5, 2, 4, 6, 8 h postdose on Days 1, 3; 2, 4h postdose on Days 2, 15; 2h postdose on Day 8; on Days 4, 5. Stage 1 Arm 2 and Stage 2, Cycle 1 of 21 days: predose (5 minutes), 0.5, 1, 1.5, 2, 4, 6h postdose on Day 2 (additionally at 8h postdose on Day 2 for Arm 2a only) ; predose (0.5h), 2h postdose on Day 9
PK-dose Proportionality as Assessed With Cmax of GDC-0575 | Stage 1 Arm 1, Cycle 1 of 21 days: predose on Days 1, 2, 3, 8, 15; postdose on Days 1, 2, 3, 4, 5, 8, 15. Stage 1 Arm 2 and Stage 2, Cycle 1 of 21 days: predose and postdose on Days 2, 9 (detailed timeframe is provided in outcome measure description)
  Stage 1 Arm 1, Cycle 1 of 21 days: predose (5 to 30 minutes) on Days 1, 2, 3, 8, 15; 0.5, 1, 1.5, 2, 4, 6, 8 h postdose on Days 1, 3; 2, 4h postdose on Days 2, 15; 2h postdose on Day 8; on Days 4, 5. Stage 1 Arm 2 and Stage 2, Cycle 1 of 21 days: predose (5 minutes), 0.5, 1, 1.5, 2, 4, 6h postdose on Day 2 (additionally at 8h postdose on Day 2 for Arm 2a only) ; predose (0.5h), 2h postdose on Day 9
PK-dose Proportionality as Assessed With AUC of GDC-0575 | Stage 1 Arm 1, Cycle 1 of 21 days: predose on Days 1, 2, 3, 8, 15; postdose on Days 1, 2, 3, 4, 5, 8, 15. Stage 1 Arm 2 and Stage 2, Cycle 1 of 21 days: predose and postdose on Days 2, 9 (detailed timeframe is provided in outcome measure description)
  Stage 1 Arm 1, Cycle 1 of 21 days: predose (5 to 30 minutes) on Days 1, 2, 3, 8, 15; 0.5, 1, 1.5, 2, 4, 6, 8 h postdose on Days 1, 3; 2, 4h postdose on Days 2, 15; 2h postdose on Day 8; on Days 4, 5. Stage 1 Arm 2 and Stage 2, Cycle 1 of 21 days: predose (5 minutes), 0.5, 1, 1.5, 2, 4, 6h postdose on Day 2 (additionally at 8h postdose on Day 2 for Arm 2a only) ; predose (0.5h), 2h postdose on Day 9
Phospho-Cyclin-Dependent Kinase 2 (pCdk2) Levels in Fresh Tumor | Stage 1 Arm 1: Screening (Day -21 to -1), Cycle 1 Day 4 (Cycle length=21 days). Stage 1 Arm 2a: Screening (Day -21 to -1), Days 3, 10 of Cycle 2. Stage1 Arm2b, Stage 2: Screening (Day -21 to -1), Day 3 of Weeks 4, 5 (Stage1 Arm2b), Weeks 1, 2 (Stage 2)
  Stage 1 Arm 1: Screening (Day -21 to -1), Cycle 1 Day 4 (Cycle length=21 days). Stage 1 Arm 2a: Screening (Day -21 to -1), Days 3 and 10 of Cycle 2. Stage 1 Arm 2b: Screening (Day -21 to -1), Day 3 of Weeks 4 and 5. Stage 2: Screening (Day -21 to -1), Day 3 of Weeks 1 and 2
Phospho-Cyclin-Dependent Kinase 2 (pCdk2) Levels in Skin Tissue | Stage 1 Arm 1: Screening (Day -21 to -1), Cycle 1 Day 4 (Cycle length=21 days). Stage 1 Arm 2a: Screening (Day -21 to -1), Days 3, 10 of Cycle 2. Stage1 Arm2b, Stage 2: Screening (Day -21 to -1), Day 3 of Weeks 4, 5 (Stage1 Arm2b), Weeks 1, 2 (Stage 2)
  Stage 1 Arm 1: Screening (Day -21 to -1), Cycle 1 Day 4 (Cycle length=21 days). Stage 1 Arm 2a: Screening (Day -21 to -1), Days 3 and 10 of Cycle 2. Stage 1 Arm 2b: Screening (Day -21 to -1), Day 3 of Weeks 4 and 5. Stage 2: Screening (Day -21 to -1), Day 3 of Weeks 1 and 2
Gamma-H2Ax (γ-H2Ax) Levels in Fresh Tumor | Stage 1 Arm 1: Screening (Day -21 to -1), Cycle 1 Day 4 (Cycle length=21 days). Stage 1 Arm 2a: Screening (Day -21 to -1), Days 3, 10 of Cycle 2. Stage1 Arm2b, Stage 2: Screening (Day -21 to -1), Day 3 of Weeks 4, 5 (Stage1 Arm2b), Weeks 1, 2 (Stage 2)
  Stage 1 Arm 1: Screening (Day -21 to -1), Cycle 1 Day 4 (Cycle length=21 days). Stage 1 Arm 2a: Screening (Day -21 to -1), Days 3 and 10 of Cycle 2. Stage 1 Arm 2b: Screening (Day -21 to -1), Day 3 of Weeks 4 and 5. Stage 2: Screening (Day -21 to -1), Day 3 of Weeks 1 and 2
Gamma-H2Ax (γ-H2Ax) Levels in Skin Tissue | Stage 1 Arm 1: Screening (Day -21 to -1), Cycle 1 Day 4 (Cycle length=21 days). Stage 1 Arm 2a: Screening (Day -21 to -1), Days 3, 10 of Cycle 2. Stage1 Arm2b, Stage 2: Screening (Day -21 to -1), Day 3 of Weeks 4, 5 (Stage1 Arm2b), Weeks 1, 2 (Stage 2)
  Stage 1 Arm 1: Screening (Day -21 to -1), Cycle 1 Day 4 (Cycle length=21 days). Stage 1 Arm 2a: Screening (Day -21 to -1), Days 3 and 10 of Cycle 2. Stage 1 Arm 2b: Screening (Day -21 to -1), Day 3 of Weeks 4 and 5. Stage 2: Screening (Day -21 to -1), Day 3 of Weeks 1 and 2

SECONDARY OUTCOMES:
Percentage of Participants With Objective Response as Determined Using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Baseline until disease progression or death (up to approximately 5 years)
Progression-Free Survival (PFS) as Determined Using RECIST v1.1 | Baseline until disease progression or death (up to approximately 5 years)
Duration of Objective Response as Determined Using RECIST v1.1 | Baseline until disease progression or death (up to approximately 5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (7):
- United States (5):
  - Yale Cancer Center, New Haven, Connecticut
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - The Sarah Cannon Research Inst, Nashville, Tennessee
- France (2):
  - Institut Bergonie; Oncologie, Bordeaux
  - Institut Gustave Roussy; Departement Oncologie Medicale, Villejuif

REFERENCES:
- [Derived] Italiano A, Infante JR, Shapiro GI, Moore KN, LoRusso PM, Hamilton E, Cousin S, Toulmonde M, Postel-Vinay S, Tolaney S, Blackwood EM, Mahrus S, Peale FV, Lu X, Moein A, Epler J, DuPree K, Tagen M, Murray ER, Schutzman JL, Lauchle JO, Hollebecque A, Soria JC. Phase I study of the checkpoint kinase 1 inhibitor GDC-0575 in combination with gemcitabine in patients with refractory solid tumors. Ann Oncol. 2018 May 1;29(5):1304-1311. doi: 10.1093/annonc/mdy076. PMID 29788155